CLINICAL TRIAL: NCT06746415
Title: The Effect of Robot-assisted Gait Training on Quadriceps Muscle Thickness, Balance and Gait Parameters in Chronic Stroke Patients
Brief Title: The Effect of Robot-assisted Gait Training in Individuals With Chronic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Guzin Kaya Aytutuldu, Assistant Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Biruni.Uni
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Chronic Stroke
Keywords: exercise; robotic gait training; balance; gait
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Gait Group (Active Comparator): Conventional walking training group will be given 20 minutes of NMES, 20 minutes of weight transfer, stretching, mobilization, bobath exercises and 20 minutes of parallel bar walking exercises.Patients in both groups will be treated 3 days a week, 1 hour a day for 6 weeks.
  Interventions: Other: Conventional Gait Training
- Robotic Gait Group (Experimental): . The robot-assisted walking group will receive 20 minutes of NMES, 20 minutes of weight transfer, stretching,mobilization, bobath exercises and 20 minutes of robot-assisted walking exercises. Patients in both groups will be treated 3 days a week, 1 hour a day for 6 weeks.
  Interventions: Other: Robotic Gait Training

INTERVENTIONS:
Other: Conventional Gait Training — onventional walking training group will be given 20 minutes of NMES, 20 minutes of weight transfer, stretching, mobilization, bobath exercises and 20 minutes of parallel bar walking exercises. Patients in both groups will be treated 3 days a week, 1 hour a day for 6 weeks.
  Arms: Conventional Gait Group
Other: Robotic Gait Training — The robot-assisted walking group will receive 20 minutes of NMES, 20 minutes of weight transfer, stretching,mobilization, bobath exercises and 20 minutes of robot-assisted walking exercises. Patients in both groups will be treated 3 days a week, 1 hour a day for 6 weeks
  Arms: Robotic Gait Group

SUMMARY:
The aim of our study was to investigate the effect of robot-assisted gait training on quadriceps muscle thickness, balance and gait parameters in individuals with chronic stroke.

For these purposes:-Improving gait and balance functions of patients with chronic stroke,-Increasing functional independence in daily life with walking trainings-Increase lower extremity muscle thickness with walking training, To investigate the effects of robot-assisted gait training on quadriceps muscle thickness, balance and gait parameters in individuals with chronic stroke.-It is aimed to contribute to the literature in this field by transforming the results to be obtained as a result of the study into a scientific publication

DETAILED DESCRIPTION:
The aim of this study was to investigate the effect of robot-assisted gait training on quadriceps muscle thickness, balance and gait parameters in individuals with chronic stroke.

Stroke refers to a neurological disorder caused by cerebrovascular damage. It is defined as a sudden brain attack that causes partial or complete brain dysfunction due to blockage or rupture of blood vessels of the brain. The primary symptom of stroke is hemiparesis. In addition, stroke negatively affects senses, motor function, perception, cognition and language, depending on location, etiology and infarct volume. One study reported that 85% of stroke patients had hemiparesis and more than 69% had upper limb dysfunction. Balance and gait disturbances are closely related in chronic stroke patients; balance is an İmportant determinant of walking ability and motor function. Impairments in the strength and standing balance of the paretic lower limb are consistently associated with gait performance. Changes in segmental transverse range of motion and coordination are associated with poor gait and balance abilities [5]. Research has shown a continuous relationship between quadriceps muscle thickness and gait parameters in chronic stroke patients. Sánchez-Sánchez (2019) found that reduced quadriceps muscle thickness was associated with a lower ability to produce maximal force and postural instability, especially in those with limited mobility in the community. It was showed that fewer muscle modules, which may be indicative of reduced muscle thickness, were associated with poorer gait quality. A study found that decreased quadriceps muscle thickness and increased intramuscular fat were associated with decreased gait independence.These findings suggest that maintaining or improving quadriceps muscle thickness may be important in improving gait performance in chronic stroke patients. Robot-assisted gait training has been frequently used in research in recent years and positive improvements in gait speed and stride length have been obtained. In some studies, it has been shown that there is no significant difference in gait compared to traditional treatment, only improving clinical scales more . In contrast, Aprile (2017) found that both robotic and traditional gait training improved clinical scales, but only the robotic group showed higher percentage changes in certain scales.However, no significant difference was found in gait analysis. Ronchi (2015) also showed no additional gains in gait rehabilitation with robotic therapy compared to conventional treatment.Therefore, although robotic gait training offers some benefits, more research is needed to determine the different or similar effects on balance, gait and lower extremity muscle thickness compared to traditional methods. The aim of our study was to investigate the effect of robot-assisted gait training on quadriceps muscle thickness, balance and gait parameters in individuals with chronic stroke. The following hypotheses will be examined in the study. H0: Robot-assisted gait training has no effect on quadriceps muscle thickness, balance and gait parameters in individuals with chronic stroke. H1: Robot-assisted gait training has an effect on quadriceps muscle thickness, balance and gait parameters in individuals with chronic stroke

ELIGIBILITY:
Inclusion Criteria:

* a history of cerebrovascular accident at least 6 months ago;
* a score of at least 20 on the mini mental test;
* no botulinum toxin treatment for the last 3 months;
* a score of 2 or above on the Functional Ambulation Scale;
* a score of 3 or above on the Brunnstrom motor staging scale in terms of lower extremity recovery level

Exclusion Criteria:

* presence of concomitant neurologic, orthopedic, cardiovascular disease and acute comorbidities
* severe spasticity of lower extremity muscles, more than 2 on the Modified Ashworth Scale

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Fugl Meyer Lower Extremity Assessment: | 15 minutes
  In this scale, reflexes, synergy-dependent or independent voluntary movement, coordination and speed are evaluated, with each item scoring Yazım alanları gerektiği kadar uzatılabilir 2 points. 0: Cannot complete movement/No active movement. 1: Partial movement. 2: Movement is completed/movements can be performed normally. The lowest clinically significant score in the Fugl-Meyer test is considered to be 6
Ten meter walk test | 5 minutes
  For this test, a 16-meter walking track is created with starting and ending points and the test is completed without considering the first 3 and last 3 meters of this track. When the patient starts walking, the stopwatch is started after the first three meters and the stopwatch is stopped at the end of the tenth meter. After the patient walks the last 3 meters, walking is terminated. The completion time of the test is recorded in seconds
Berg Balance Scale | 15 minutes
  The Berg Balance Scale (BBS) is a scale that includes 14 instructions and for each instruction, the patient's performance is observed and a score between 0-4 is given.
  A score of 0 is given when the patient cannot perform the activity at all, while a score of 4 is given when the patient completes the activity independently. The highest score is 56, with 0-20 points indicating impaired balance, 21-40 points indicating acceptable balance, and 41-56 points indicating good balance. The scale takes between 10 and 20 minutes to complete.
  It has been validated in patients with chronic stroke
Examination of muscle thickness by ultrasound | 10 minutes
  The muscle thickness of the quadriceps and tibialis anterior muscles on the hemiplegic and intact side will be measured and recorded by ultrasound before and after treatment.
Gait Analysis with Kinovea | 10 minutes
  Walking distances of 3 meters will be recorded with the camera to be placed on the sagittal. Colored marks will be placed on the right and left heels.
  The colored marks will be marked on the video and step lengths, walking speed and arm swing will be calculated with Kinovea motion analysis software. Several gait cycles will be recorded in the video and cadence (number of steps per minute), right and left step lengths will be expressed

SECONDARY OUTCOMES:
The Timed Up and Go Test | 5 minutes
  The Timed Up and Go Test is a simple, widely used and quick test to assess mobility, balance and fall risk. To perform the test, participants need to get up from a standard chair, walk comfortably to a location 3 meters away from the floor, turn around, walk back to the chair and sit down in the same chair. All steps of the test will be measured using a stopwatch
Stroke Specific Quality of Life Scale | 15 minutes
  This scale, which was created to assess the quality of life of people diagnosed with stroke, consists of 12 domains including 49 items and is scored with a five-point Likert scale. In determining the mean score of each domain of the scale, the scores obtained from all items belonging to the domain are summed and divided by the number of items belonging to the domain. The total score of the scale is calculated by dividing the sum of the average scores obtained from each domain by 12. A high scale score indicates a high quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Güzin Kaya Aytutuldu, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang JJ, Tung WL, Wu WL, Su FC. Effect of bilateral reaching on affected arm motor control in stroke--with and without loading on unaffected arm. Disabil Rehabil. 2006 Dec 30;28(24):1507-16. doi: 10.1080/09638280600646060. PMID 17178614
- [Background] Yoo DH, Kim SY. Effects of upper limb robot-assisted therapy in the rehabilitation of stroke patients. J Phys Ther Sci. 2015 Mar;27(3):677-9. doi: 10.1589/jpts.27.677. Epub 2015 Mar 31. PMID 25931706
- [Background] Lee KB, Lim SH, Kim YD, Yang BI, Kim KH, Lee KS, Kim EJ, Hwang BY. The contributions of balance to gait capacity and motor function in chronic stroke. J Phys Ther Sci. 2016 Jun;28(6):1686-90. doi: 10.1589/jpts.28.1686. Epub 2016 Jun 28. PMID 27390395
- [Background] Hacmon RR, Krasovsky T, Lamontagne A, Levin MF. Deficits in intersegmental trunk coordination during walking are related to clinical balance and gait function in chronic stroke. J Neurol Phys Ther. 2012 Dec;36(4):173-81. doi: 10.1097/NPT.0b013e31827374c1. PMID 23095903
- [Background] Sanchez-Sanchez ML, Ruescas-Nicolau MA, Carrasco JJ, Espi-Lopez GV, Perez-Alenda S. Cross-sectional study of quadriceps properties and postural stability in patients with chronic stroke and limited vs. non-limited community ambulation. Top Stroke Rehabil. 2019 Oct;26(7):503-510. doi: 10.1080/10749357.2019.1634360. Epub 2019 Jun 27. PMID 31246150
- [Background] Shin J, An H, Yang S, Park C, Lee Y, You SJH. Comparative effects of passive and active mode robot-assisted gait training on brain and muscular activities in sub-acute and chronic stroke. NeuroRehabilitation. 2022;51(1):51-63. doi: 10.3233/NRE-210304. PMID 35311717